CLINICAL TRIAL: NCT06487793
Title: A Mobile App to Address Co-Occurring Sleep Problems and Heavy Alcohol Use Among Veterans Outside of Care Settings
Brief Title: Mobile App Intervention for Sleep Problems and Alcohol Use Among Veterans
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: RAND (Other); Palo Alto Veterans Institute for Research (Other); University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Eric Pedersen, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34AA030868 (NIH)
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Alcohol Use Disorder; Insomnia
MeSH Terms: conditions — Alcoholism; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are asked to complete one of two mobile phone-based programs. They may not know which condition is the experimental condition and which is the control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Insomnia Coach Mobile App Intervention (Experimental): Participants assigned to the experimental condition are asked to view the modules within the app for 8 weeks. The mobile app contains content based on cognitive behavioral therapy for insomnia (CBT-I) enhanced with content from brief alcohol interventions.
  Interventions: Behavioral: Enhanced Insomnia Coach
- Sleep Hygiene Control (Active Comparator): Participants assigned to the control condition are asked to view sleep hygiene modules delivered by email once per week for 8 weeks.
  Interventions: Behavioral: Sleep hygiene comparator

INTERVENTIONS:
Behavioral: Enhanced Insomnia Coach — The intervention combines the Insomnia Coach app with additional brief alcohol intervention to facilitate behavior change for both drinking behavior and insomnia symptoms. Insomnia Coach contains multiple components of CBT-I (e.g., stimulus control, cognitive restructuring, relaxation training, sleep hygiene/psychoeducation, monitoring of sleep via journals). The brief alcohol intervention content added to the CBT-I app is based on CBT skills for moderate drinking, delivered in a motivational enhancement style, and has demonstrated efficacy among young adults and veterans (e.g., correcting perceived norms, use of protective behavioral strategies, challenging expectancies).
  Arms: Enhanced Insomnia Coach Mobile App Intervention
Behavioral: Sleep hygiene comparator — Content is based on sleep hygiene practices, but without additional CBT-I content featured in the experimental condition. There is also not brief alcohol intervention content in the control condition.
  Arms: Sleep Hygiene Control

SUMMARY:
The goal of this clinical trial is to test the preliminary efficacy of a brief mobile app targeting insomnia symptoms among veterans. In this study, we will enhance the mobile app, Insomnia Coach, with content from brief alcohol interventions to help veterans reduce both insomnia symptoms and alcohol use behaviors. We will compare those veterans who are randomly assigned to receive this brief mobile app intervention to those who receive a control condition. This will help us determine if veterans randomly assigned to receive the intervention experience greater improvement on outcomes compared to those who do not receive the intervention. The study involves a beta-test phase of the app to ensure feasibility and acceptability by veterans, followed by a randomized controlled trial with 130 veterans who meet criteria for insomnia and alcohol use disorder.

ELIGIBILITY:
Inclusion Criteria:

* U.S. veteran aged 18 or older separated or discharged from service in the Air Force, Army, Marine Corps, Navy, or Coast Guard
* Not currently affiliated with active duty service or on active reserves or guard service
* Served since September 11, 2001
* No past 6-month treatment for alcohol or drug use or insomnia
* Alcohol Use Disorder Identification Test (AUDIT) score of 8 or higher
* Insomnia Severity Index (ISI) score of 10 or higher

Exclusion Criteria:

* Positive screening for other substance use disorders (not including cannabis use disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia symptoms | Past 30 days
  7-item Insomnia Severity Index (ISI). The ISI is a measure of insomnia symptoms including difficulty falling/staying asleep, sleep problems interfering with daily life, and concern about sleep problems.
Alcohol use frequency | Past 30 days
  Days used in past 30 days
Alcohol use quantity | Past 30 days
  Number of drinks per drinking occasion

SECONDARY OUTCOMES:
Sleep quality | Past 30 days
  The 19-item Pittsburgh Sleep Quality Index will assess nuanced sleep behaviors at each time point (e.g., sleep latency, sleep duration, subjective sleep quality)
Alcohol-related consequences | Past 30 days
  15-item Short Inventory of Alcohol Problems assesses problems from alcohol use across multiple domains such as interpersonal, intrapersonal, and physical.

OTHER OUTCOMES:
Treatment initiation | Past 30 days
  Affirmative responses regarding whether participants initiated more formal treatment since starting the study

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared in accordance with NIH guidelines and uploaded to the NDA repository.